CLINICAL TRIAL: NCT03694041
Title: Double Blind, Randomized Study Assessing the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses or Multiple Ascending Doses of APX-115 in Healthy Male Volunteers.
Brief Title: Safety, Tolerability, PK and PD of SAD or MAD of APX-115 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP101817.APT; 2017-004252-30 (EudraCT Number)
Record Dates: First submitted 2018-09-20; First posted 2018-10-03 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Healthy; Safety
MeSH Terms: interventions — isuzinaxib

STUDY DESIGN:
Intervention Model Description: Parallel design for SAD and MAD studies Crossover design for Food and Drug interaction studies
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- SAD: APX-115 (Experimental): Experimental: APX-115 SAD group
  Interventions: Drug: SAD: APX-115
- SAD: Placebo (Placebo Comparator): Experimental: Placebo group
  Interventions: Drug: SAD: Placebo
- MAD: APX-115 (Experimental): Experimental: APX-115 MAD group
  Interventions: Drug: MAD: APX-115
- MAD: Placebo (Placebo Comparator): Experimental: Placebo group
  Interventions: Drug: MAD: Placebo
- Food effect - Fasting condition (Active Comparator): Experimental: APX-115 under fasting condition
  Interventions: Other: Food effect: fasted and fed
- Food effect - fed condition (Active Comparator): Experimental: APX-115 under fed condition
  Interventions: Other: Food effect: fasted and fed
- Drug Interaction - metabolic probe (Placebo Comparator): Experimental: metabolic probe
  Interventions: Other: Metabolic probe with or without APX-115

INTERVENTIONS:
Drug: SAD: APX-115 — Drug: APX-115 SAD APX-115 SAD for 1day
  Arms: SAD: APX-115
Drug: SAD: Placebo — Drug: Placebo Placebo for 1day
  Arms: SAD: Placebo
Drug: MAD: APX-115 — Drug: APX-115 MAD APX-115 MAD repeatedly administered.
  Arms: MAD: APX-115
Drug: MAD: Placebo — Matching study drug will be repeatedly administered.
  Arms: MAD: Placebo
Other: Food effect: fasted and fed — A single dose of APX-115, selected from the SAD study, will be administered under fasted and fed condition.
  Arms: Food effect - Fasting condition; Food effect - fed condition
Other: Metabolic probe with or without APX-115 — A metabolic probe will be administered with and without APX-115.
  Arms: Drug Interaction - metabolic probe

SUMMARY:
This study aims to evaluate the safety, tolerabilty, pharmacokinetics and pharmacodynamics of single ascending doses and multiple ascending doses of APX-115 in healthy males. This study also aims to evaluate the effect of food consumption on the pharmacokinetics of APX-115 and potential interaction between caffeine and APX-115 in healthy males.

ELIGIBILITY:
Inclusion:

* Healthy male subject, aged between 18 and 45 years inclusive
* Certified as healthy by a comprehensive clinical assessment
* Normal dietary habits
* Normal ECG recording on a 12-lead ECG
* Signing a written informed consent prior to selection

Exclusion:

* Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic, infectious or ocular disease
* Frequent headaches and / or migraine, recurrent nausea and / or vomiting
* Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position
* Blood donation (including in the frame of a clinical trial) within 2 months before administration
* General anaesthesia within 3 months before administration
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician
* Inability to abstain from intensive muscular effort
* No possibility of contact in case of emergency
* Any drug intake (except paracetamol or contraception) during the last month prior to the first administration
* History or presence of drug or alcohol abuse (alcohol consumption > 30 grams / day)
* Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day)
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
* Positive results of screening for drugs of abuse
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
* Administrative or legal supervision

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
SAD: incidence of treatment emergent adverse events | Up to Day 8
SAD: number of clinically significant abnormal findings from vital signs (blood pressure, pulse) | Up to Day 8
SAD: number of clinically significant abnormal findings from physical exam | Up to Day 8
SAD: number of clinically significant abnormal findings from electrocardiogram | Up to Day 8
SAD: number of clinically significant abnormal findings from biological tests | Up to Day 8
MAD: incidence of treatment emergent adverse events | Up to Day 17
MAD: number of clinically significant abnormal findings from vital signs (blood pressure, pulse) | Up to Day 17
MAD: number of clinically significant abnormal findings from physical exams | Up to Day 17
MAD: number of clinically significant abnormal findings from electrocardiogram | Up to Day 17
Food effect: peak serum concentration (Cmax) of APX-115 under fasting and fed conditions | Up to Day 4 post-dose
Food effect: time to reach the Cmax (Tmax) of APX-115 under fasting and fed conditions | Up to Day 4 post-dose
Food effect: area under the curve (AUC) of APX-115 under fasting and fed conditions | Up to Day 4 post-dose
Food effect: elimination rate constant (Kel) of APX-115 under fasting and fed conditions | Up to Day 4 post-dose
Food effect: ratio AUCfed/AUCfasted | Up to Day 4 post-dose
Drug interaction: peak serum concentration (Cmax) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: Time to reach the Cmax (tmax) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction study: Area under the Curve (AUC) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: elimination rate constant (Kel) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: half-life (t1/2) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: volume of distribution (Vd/f) of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: clearance of a metabolic probe or APX-115 | Up to Day 4 post-dose
Drug interaction: Incidences of treatment emergent adverse events | Up to Day 4 post-dose

SECONDARY OUTCOMES:
SAD: time to reach Cmax (Tmax) of APX-115 | Up to Day 5
SAD: peak serum concentration (Cmax) of APX-115 | Up to Day 5
SAD: lowest plasma concentration before next dosing (Ctrough) | Up to Day 5
SAD: Area Under the Curve (AUC) of APX-115 | Up to Day 5
SAD: volume of distribution (Vd/F) of APX-115 | Up to Day 5
SAD: clearance (CL/F) of APX-115 | Up to Day 5
MAD: peak serum concentration (Cmax) of APX-115 | Up to Day 11
MAD: time to reach the Cmax (Tmax) of APX-115 | Up to Day 11
MAD: Area Under the Curve (AUC) of APX-115 | Up to Day 11
MAD: lowest plasma concentration of APX-115 before next dosing (Ctrough) | Up to Day 11
MAD: volume of distribution (Vd/F) of APX-115 | Up to Day 11
MAD: Clearance (CL/F) of APX-115 | Up to Day 11
MAD: accumulation ratio | Up to Day 11
Food effect & drug interaction: incidence of treatment emergent adverse events | Up to Day 4 post-dose
Food effect & drug interaction: number of clinically significant findings from vital signs (blood pressure and pulse) | Up to Day 4 post-dose
Food effect & drug interaction: number of clinically significant findings from physical exam | Up to Day 4 post-dose
Food effect & drug interaction: number of clinically significant findings from electrocardiogram | Up to Day 4 post-dose
Food effect & drug interaction: number of clinically significant findings from biological tests | Up to Day 4 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: Undecided